CLINICAL TRIAL: NCT04687358
Title: Registry of the Natural History of Recurrent Pericarditis in Pediatric and Adult Patients
Acronym: RESONANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Kiniksa Pharmaceuticals International, plc (Industry)
Collaborators: Kiniksa Pharmaceuticals (UK), Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KPL-914-Reg-001
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active RP: Patients who are currently under the care of a physician for treatment of RP, currently on treatment for RP, and have had an episode (recurrence of typical pericarditis pain associated with supportive objective evidence of pericarditis) in the last 3 years prior to enrollment. Once included in the registry, these patients will have both retrospective and prospective follow-up and data collection (hybrid design).
- Inactive RP: Patients who have had a diagnosis of RP, have not had an episode for 3 years and have not been prescribed any treatment for RP in the last 3 years, prior to enrolling in the registry. Once included in the registry, data collected from these patients will be retrospective only.

SUMMARY:
The registry will focus on furthering the understanding of the natural history of recurrent pericarditis (RP), as well as document RP-related clinical, health-related quality of life (HRQoL), and economic burden and will assist the medical community to refine or develop data-driven recommendations for clinical management of RP patients to optimize clinical outcomes. It also aims to generate data in support of the impact of rilonacept on clinical outcomes in a real-world population.

ELIGIBILITY:
ACTIVE RP PATIENTS

Select Inclusion Criteria:

* Physician-confirmed (or confirmation in medical records) diagnosis of RP defined as an initial, acute, episode and at least one pericarditis recurrence after the initial acute episode
* Experienced at least one pericarditis episode in the 3 years prior to inclusion
* Under the care of a physician for the treatment and management of RP
* Currently prescribed medication for RP

Select Exclusion Criteria:

* Diagnosis of pericarditis secondary to tuberculosis (TB), cancer if not in full remission, post thoracic blunt trauma (e.g., motor-vehicle accidents), myocarditis, systemic autoimmune diseases, except SJIA and adult Still's disease, HIV
* Appears to have an impairment (e.g., cognitive, hearing, visual) or insufficient English or Spanish proficiency that could interfere with ability to complete patient-completed assessments
* Currently enrolled in a therapeutic investigational drug or device study

INACTIVE RP PATIENTS

Select Inclusion Criteria:

* Physician-confirmed (or confirmation in medical records) diagnosis of RP defined as an initial, acute, episode and at least one pericarditis recurrence after the initial, acute episode
* Patient had a last episode occurring at least 3 years and up to 5 years before registry inclusion
* Resolution of RP symptoms confirmed with no further RP treatment for 3 years prior to registry enrollment

Select Exclusion Criteria:

* Experienced a pericarditis episode within 3 years from enrolling in the registry
* Currently receiving RP treatment prescribed by a treating physician (e.g., CS, colchicine)
* Diagnosis of pericarditis secondary to tuberculosis (TB), cancer if not in full remission, post thoracic blunt trauma (e.g., motor-vehicle accidents), myocarditis, systemic autoimmune diseases except SJIA and adult Still's disease, HIV
* Enrolled in a therapeutic investigational clinical trial during the observation period

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with active or inactive recurrent pericarditis who have participated in the RHAPSODY (KPL-914-C002) Phase 3 clinical study of rilonacept and patients from sites who have expressed an interest in the registry will be included. In addition, RESONANCE will also include decentralized sites for remote patients who wish to participate in the registry but are not near a registry site.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patients using 1 or more RP treatments | 5 years
  Proportion of patients using 1, 2, 3, or more concomitant RP treatments

SECONDARY OUTCOMES:
Most frequently used RP treatments | 5 years
  Number of subjects who used each treatment recorded during the study
Reduction in the use of corticosteroids | 5 years
  Change from baseline through end of observation in corticosteroid use
Change in RP activity | 1 year
  Change from baseline in RP disease recurrences within 1 year (from 1 year prior to baseline to 1 year after baseline
Change in pericardial rub | 5 years
  Change from baseline in pericardial rub
Change in pericardial effusion | 5 years
  Change from baseline in pericardial effusion
Change in fever | 5 years
  Change from baseline in fever
Change in dyspnea | 5 years
  Change from baseline in dyspnea
Change in C-reactive protein (CRP) | 5 years
  Change from baseline in CRP
Change in erythrocyte sedimentation rate (ESR) | 5 years
  Change from baseline in ESR
Change in white blood count (WBC) | 5 years
  Change from baseline in WBC
Change in interleukin-1 (IL-1) | 5 years
  Change from baseline in IL-1
Change in interleukin-6 (IL-6) | 5 years
  Change from baseline in IL-6
Change in electrocardiogram (ECG) | 5 years
  Change from baseline in ST-, PR-, QRS- and QT- intervals
Change in echocardiogram | 5 years
  Change from baseline in echocardiogram
Change in chest x-ray | 5 years
  Change from baseline in chest x-ray
Change in cardiac magnetic resonance imaging (cMRI) | 5 years
  Change from baseline in cMRI
Change in cardiovascular magnetic resonance (CMR) imaging | 5 years
  Change from baseline in CMR
Change in Multidetector (cardiac) computed tomography (MDCT) | 5 years
  Change from baseline in MDCT
Adverse event rate | 5 years
  Rate of adverse events reported by PC treatment
Changes in PROMIS-29 patient-reported outcomes | 5 years
  Change from baseline in PROMIS-29
Changes in PROMIS Pediatric/Parent 25 patient-reported outcomes | 5 years
  Change from baseline in PROMIS Pediatric/Parent 25
Changes in insomnia severity index (ISI) patient-reported outcomes | 5 years
  Change from baseline in ISI
Changes in Patient Global Impression of Pericarditis Severity (PGIPS) patient-reported outcomes | 5 years
  Change from baseline in PGIPS
Changes in persistent pericarditis numerical rating scale (PPNRS) patient-reported outcomes | 5 years
  Change from baseline in PPNRS
Changes in D12 patient-reported outcomes | 5 years
  Change from baseline in D12 outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: John F Paolini, MD, PhD, Study Director — Kiniksa Pharmaceuticals Corp
Locations (29):
- United States (29):
  - Alaska Heart & Vascular Institute, Anchorage, Alaska
  - Pima Heart and Vascular, Tucson, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Scripps Health, San Diego, California
  - Northwestern University, Chicago, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Barnes-Jewish Hospital/Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - TKL Research Inc., Fair Lawn, New Jersey
  - NYU Langone Health, New York, New York
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - The Linder Research Center at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Legacy Medical Group, Cardiology, Portland, Oregon
  - Carnegie Mellon University, Allegheny Health Network, Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center - Cherry Hill, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided